CLINICAL TRIAL: NCT04202315
Title: Use of Virtual Reality for Pelvic External Fixator Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Reza Firoozabadi, Associate Professor, School of Medicine: Orthopaedics and Sports Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002673
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Pelvic Fracture Pubic Rami Multiple - Unstable Closed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care, no Virtual Reality
- Virtual Reality (Experimental): Standard of care plus Virtual Reality
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Utilizing Virtual Reality during external fixator removal in outpatient clinic setting.
  Arms: Virtual Reality

SUMMARY:
Assessing the role of virtual reality in decreasing pain and improving patient satisfaction in outpatient removal of pelvic external fixator constructs.

ELIGIBILITY:
Inclusion Criteria:

* Pelvis external fixator placed at study institution
* External fixator placed for pelvic instability

Exclusion Criteria:

* Infected pin or pins
* Loose pin or pins
* Psych history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | During procedure
  Pain score during removal of external fixator

SECONDARY OUTCOMES:
Patient Satisfaction | immediately after procedure
  Self reported patient satisfaction, comparing no virtual reality to virtual reality

CONTACTS AND LOCATIONS:
Overall Officials: Reza Firoozabadi, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington/Harborview Medical Center, Seattle, Washington, United States